CLINICAL TRIAL: NCT07341919
Title: Subtenon Autologous Platelet-Rich Plasma in Inherited and Degenerative Retinal Diseases: A Prospective Comparative Pilot Study
Brief Title: Subtenon Autologous Platelet-Rich Plasma in Inherited and Degenerative Retinal Diseases
Acronym: RETINA-PRP
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rubens Camargo Siqueira (Other)
Responsible Party: Sponsor-Investigator, Rubens Camargo Siqueira, MD,PhD, Centro de Pesquisa Rubens Siqueira
Organization: Centro de Pesquisa Rubens Siqueira (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RETINA-PRP Study
Record Dates: First submitted 2025-12-13; First posted 2026-01-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Extensive Macular Atrophy With Pseudodrusen (EMAP); Retinitis Pigmentosa (RP)
Keywords: Retinitis pigmentosa; EMAP; Macular Atrophy; Pseudodrusen-like; platelet-rich plasma; PRP
MeSH Terms: conditions — Retinitis Pigmentosa; Anetoderma

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, open-label interventional pilot study designed to assess the ocular safety, feasibility, and functional outcomes of subtenon administration of autologous platelet-rich plasma (PRP) in patients with degenerative retinal diseases.
  All participants receive three subtenon injections of autologous PRP (1.5 mL per injection) administered at baseline (M0) and at two-month intervals (M2, M4).
  Given the exploratory nature of the study and the heterogeneity of degenerative retinal diseases, no randomization or masking is applied. Each participant serves as their own control, with outcomes evaluated as within-subject changes from baseline to six months (M0-M6).
  The study aims to provide proof-of-concept data on the regenerative and immunomodulatory potential of PRP, focusing on functional outcomes and OCT-based biomarkers, to support the design of future controlled trials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subtenon Injection of Autologous Platelet-Rich Plasma (Experimental): Experimental: Subtenon Injection of Autologous Platelet-Rich Plasma Participants receive subtenon injections of autologous platelet-rich plasma (PRP), 1.5 mL per injection, administered at baseline (M0), month 2 (M2), and month 4 (M4).
  This arm evaluates the effect of local autologous regenerative and immunomodulatory therapy on visual function and retinal structure in patients with degenerative retinal diseases, including Retinitis Pigmentosa and Extensive Macular Atrophy with Pseudodrusen-like Appearance (EMAP).
  Interventions: Biological: Subtenon Injection of Autologous Platelet-Rich Plasma

INTERVENTIONS:
Biological: Subtenon Injection of Autologous Platelet-Rich Plasma — Biological: Subtenon Autologous Platelet-Rich Plasma Participants receive subtenon injections of autologous platelet-rich plasma (PRP), 1.5 mL per injection, administered at baseline (M0), month 2 (M2), and month 4 (M4).
  Other Names: PRP

SUMMARY:
his prospective, comparative pilot study investigates the safety and functional outcomes of subtenon autologous platelet-rich plasma (PRP) in patients with Retinitis Pigmentosa (RP) and Extensive Macular Atrophy with Pseudodrusen-like Appearance (EMAP).

Participants will receive three subtenon injections of autologous platelet-rich plasma (1.5 mL per injection) administered at two-month intervals (M0, M2, M4).

The primary objective is to assess functional changes over a 6-month period, with a focus on visual field preservation, evaluated by the Field Preservation Deviation Index (FPDI) and Mean Deviation (MD), as well as best-corrected visual acuity (BCVA, LogMAR).

Secondary outcomes include changes in 30-Hz flicker electroretinography (ERG) amplitude, structural retinal parameters on optical coherence tomography (OCT)-including central macular thickness and ellipsoid zone length-and ocular safety outcomes, such as intraocular pressure, local tolerability, and the occurrence of inflammatory or adverse events related to subtenon PRP administration.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a genetically and phenotypically heterogeneous group of inherited retinal dystrophies characterized by progressive degeneration of photoreceptors, typically initiating with rod dysfunction and followed by secondary cone involvement. This process leads to nyctalopia, progressive constriction of the visual field, and, in advanced stages, impairment of central vision. Although recent advances in gene-specific and cell-based therapies have expanded treatment possibilities for selected subgroups, the majority of patients with RP still lack broadly applicable therapeutic approaches capable of modifying disease progression.

Extensive Macular Atrophy with Pseudodrusen-like Appearance (EMAP) is a distinct degenerative macular phenotype characterized by early-onset bilateral macular atrophy associated with pseudodrusen-like deposits, progressive loss of the outer retina and retinal pigment epithelium, and marked chorioretinal thinning. Despite its phenotypic differences from classical inherited retinal dystrophies, EMAP shares several pathobiological mechanisms with RP, including photoreceptor degeneration, outer retinal ischemia, chronic para-inflammatory activity, microglial activation, and progressive macular atrophy, ultimately resulting in severe central vision loss.

Accumulating experimental and clinical evidence suggests that both RP and EMAP are driven not only by primary degenerative mechanisms but also by sustained para-inflammatory processes at the level of the outer retina, retinal pigment epithelium, and choroid. Dysregulation of microglial activity, oxidative stress, complement activation, and chronic release of inflammatory mediators may contribute to secondary neuronal damage and accelerate structural and functional decline. These shared biological pathways provide a rationale for exploring therapeutic strategies with combined neurotrophic, anti-inflammatory, and tissue-supportive effects.

Autologous platelet-rich plasma (PRP) has emerged as a potential multimodal biologic therapy due to its high concentration of endogenous growth factors and cytokines, including platelet-derived growth factor, transforming growth factor-beta, insulin-like growth factor-1, basic fibroblast growth factor, and other bioactive mediators. These factors may support retinal homeostasis by modulating inflammatory signaling, enhancing chorioretinal perfusion, and promoting cellular survival pathways within the neuroretina and retinal pigment epithelium.

The subtenon route of administration was selected to enable gradual diffusion of PRP-derived bioactive factors toward the posterior segment while minimizing risks associated with intravitreal delivery. This approach is particularly suited for chronic degenerative retinal diseases, where safety, repeatability, and long-term tolerability are essential considerations.

This prospective pilot study was designed to assess the feasibility and ocular safety of repeated subtenon administration of autologous PRP in patients with RP and EMAP, while exploring functional and structural signals over a defined follow-up period. By integrating multimodal functional and imaging assessments, the study aims to generate preliminary data to inform the design of future controlled clinical trials evaluating regenerative and immunomodulatory strategies for inherited and degenerative retinal disorders characterized by progressive photoreceptor loss and macular atrophy.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Clinical diagnosis of retinitis pigmentosa (RP) or EMAP (Extensive Macular Atrophy with Pseudodrusen-like Appearance), confirmed by multimodal evaluation.
* Best-corrected visual acuity (BCVA) ≥ counting fingers at 1 meter (approximately ≤ 1.9 logMAR) in the study eye.
* Measurable visual field on iCare COMPASS (10-2 or 24-2) with acceptable reliability indices.
* Clear ocular media adequate for safe intravitreal injection and high-quality optical coherence tomography (OCT) imaging.
* Ability and willingness to provide written informed consent.
* Ability to comply with scheduled study visits, including:

  * Baseline (M0)
  * Day 7-14 after injections
  * Month 2 (M2), Day 7-14
  * Month 4 (M4), Day 7-14
  * Month 6 (M6)
* For ERG subset only:

  o Presence of a recordable baseline 30-Hz flicker electroretinogram (ERG) response, defined as a signal-to-noise ratio ≥ 3:1 and amplitude ≥ 3.0 μV.
* Note: Absence of a measurable flicker ERG response does not exclude participation in the main study.

Exclusion Criteria

* Active ocular inflammation (anterior, intermediate, or posterior uveitis) or active infectious ocular disease in the study eye.
* Active choroidal neovascularization or other macular diseases unrelated to RP or EMAP.
* Uncontrolled glaucoma (intraocular pressure > 21 mmHg despite therapy) or optic neuropathies not related to RP or EMAP.
* Significant media opacity that may impair imaging quality or compromise the safety of intravitreal injection.
* Recent ocular interventions that may confound study outcomes, including:

  * Intravitreal therapy within 3 months prior to enrollment.
  * Periocular corticosteroid injection within 3 months prior to enrollment.
  * Major intraocular surgery within 3 months prior to enrollment.
* Known hypersensitivity to adalimumab, povidone-iodine, local anesthetics, or any component of the study formulations.
* Coagulopathy or contraindications to ocular injections, including:

  * Platelet count < 100,000/μL, or
  * INR > 1.5 unless adequately corrected.
* Pregnancy or breastfeeding.
* Women of childbearing potential unwilling to use effective contraception during the study period.
* Uncontrolled systemic disease that, in the investigator's judgment, increases risk or interferes with study participation or completion.
* Participation in another interventional clinical trial within 3 months prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-04 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Change in Field Preservation Deviation Index (FPDI) | Baseline to Month 6
  Change (Δ) in Field Preservation Deviation Index (FPDI), expressed as a percentage (%), measured by automated perimetry using the iCare COMPASS system. The FPDI reflects the proportion of preserved visual field relative to age-matched normative data and provides a quantitative assessment of global visual field integrity. The outcome is defined as the difference between baseline (Month 0) and Month 6 values in the study eye.
. Change in Mean Deviation (MD) | Baseline to Month 6
  Change (Δ) in Mean Deviation (MD), expressed in decibels (dB), measured by automated perimetry using the iCare COMPASS system. Mean Deviation represents the average difference in retinal sensitivity compared with age-adjusted normative values, serving as a global index of visual field loss. The outcome corresponds to the difference between baseline (Month 0) and Month 6 measurements in the study eye.
. Change in Best-Corrected Visual Acuity (BCVA) | Baseline to Month 6
  Change (Δ) in Best-Corrected Visual Acuity (BCVA), expressed in logarithm of the minimum angle of resolution (LogMAR), measured using standardized Early Treatment Diabetic Retinopathy Study (ETDRS) charts under controlled testing conditions. BCVA assesses central visual function and foveal integrity. The outcome is defined as the difference between baseline (Month 0) and Month 6 BCVA values in the study eye.

SECONDARY OUTCOMES:
Change in Pattern Standard Deviation (PSD) | Baseline to Month 6]
  Change (Δ) in Pattern Standard Deviation (PSD), expressed in decibels (dB), measured by automated perimetry using the iCare COMPASS system. PSD reflects localized irregularities in visual field sensitivity and is particularly sensitive to focal or non-uniform patterns of visual field loss. The outcome is defined as the difference between baseline (Month 0) and Month 6 measurements in the study eye.
Change in 30-Hz Flicker ERG Amplitude | Baseline to Month 6
  Change (Δ) in 30-Hz flicker electroretinogram (ERG) amplitude, expressed in microvolts (µV), measured in accordance with International Society for Clinical Electrophysiology of Vision (ISCEV) standards. The 30-Hz flicker ERG primarily assesses cone-mediated retinal function and provides an objective measure of global photoreceptor and post-receptoral pathway integrity. The outcome corresponds to the difference between baseline (Month 0) and Month 6 values in the study eye.
Change in Central Macular Thickness (CMT) | Baseline to Month 6
  Change (Δ) in central macular thickness (CMT), expressed in micrometers (µm), measured by spectral-domain optical coherence tomography (SD-OCT). CMT represents the average retinal thickness within the central macular subfield and serves as a structural biomarker of macular integrity, including retinal edema, atrophy, or remodeling. The outcome is defined as the difference between baseline (Month 0) and Month 6 measurements in the study eye.
Change in Ellipsoid Zone (EZ) Length | Baseline to Month 6
  Change (Δ) in ellipsoid zone (EZ) length, expressed in micrometers (µm), measured by spectral-domain optical coherence tomography (SD-OCT). EZ length reflects the integrity and spatial extent of photoreceptor inner segment ellipsoid band and is a sensitive structural biomarker of photoreceptor preservation in degenerative retinal diseases. The outcome corresponds to the difference between baseline (Month 0) and Month 6 measurements in the study eye.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens C Siqueira, MD,PhD, Principal Investigator — Rubens Siqueira Research Center
Locations (1):
- Centro Especializado Retina e Vítreo, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided